CLINICAL TRIAL: NCT04657835
Title: Multiparametric MRI Assessment of Atrial Heart Disease as a Predictor of Atrial Fibrillation After Myocardial Revascularization Surgery
Acronym: IRM-FAPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20CH027; ANSM (Other: 2026-A00173-48)
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Atrial Fibrillation
Keywords: magnetic resonance imaging; implantable holter monitor; atrial heart disease
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective single-center pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myocardial revascularization cardiac surgery by coronary artery bypass grafting (Experimental): Patient with indication of Coronary Artery Bypass Grafting will be included. They will have:
  * before surgery : 4D cardiac MRI with gadoteric acid + ILR implantation + blood sampling
  * during surgery : right atrial biopsy
  * after surgery : Continuous monitoring by ILR for 12 months + scheduled clinical consultation (at 12 months)
  Interventions: Device: 4D cardiac MRI with gadoteric acid; Biological: Blood sample; Device: Implantable Loop Recorder (ILR); Procedure: Right atrial biopsy

INTERVENTIONS:
Device: 4D cardiac MRI with gadoteric acid — 4D cardiac MRI with gadoteric acid injection will be performed prior the surgery, according to a standardized technical protocol.
  Other Names: 4D flow Magnetic Resonance Imaging with Late Gadolinium Enhancement
Biological: Blood sample — Peripheral venous blood sample (1 x 6 ml EDTA tube): taken during preoperative assessment to measure inflammatory biomarkers (CRP, IL-1, TNF-α).
Device: Implantable Loop Recorder (ILR) — Implantation of a Holter monitor (Implantable Loop Recorder) prior to surgery, performed preoperatively under local anesthesia.
  The ILR will enable continuous recording of the heart rhythm for 12 months with automatic data transmission via remote monitoring. The minimally invasive procedure will be performed by an experienced cardiologist under the usual safety conditions.
Procedure: Right atrial biopsy — During the surgical procedure (coronary artery bypass grafting), a right atrial biopsy will be performed using a brief, low-risk procedure on a small tissue sample. The sample will be analyzed using Masson's trichrome staining to assess atrial fibrosis.

SUMMARY:
Postoperative atrial fibrillation (POAF) occurs in 20-40% of patients undergoing coronary artery bypass grafting (CABG) and is a marker of atrial vulnerability. It is strongly associated with AF recurrence, stroke, and cardiovascular mortality. It presents risk factors with atrial heart disease.

The latter refers to all structural, electrical, and mechanical alterations of the atrium that create a substrate conducive to AF.

Multiparametric cardiac MRI is currently the most comprehensive test for assessing atrial heart disease, thanks to its structural and functional analysis (atrial fibrosis, atrial strain, intracavitary 4D flow). However, to date, no prospective study has evaluated these parameters as predictors of AF recurrence after CAP. At the same time, an implantable Holter monitor will be used to enable detailed and continuous detection of recurrence episodes, overcoming the limitations of conventional monitoring strategies. By combining multiparametric imaging, histological analysis, and continuous monitoring for the first time, this study proposes a paradigm shift in the assessment of postoperative AF: moving from a descriptive and ad hoc approach to a mechanistic, integrative, and predictive approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for surgical myocardial revascularization by isolated coronary artery bypass grafting, to be performed in the cardiac surgery department of Saint-Étienne University Hospital.
* Patient affiliated with or entitled to social security coverage
* Patient who has received informed information about the study and has co-signed, with the investigator, a consent form to participate in the study

Exclusion Criteria:

* Contraindication related to cardiac MRI
* Contraindication related to ILR implantation
* Documented history of atrial fibrillation
* Concomitant indication for valve surgery or other associated cardiac intervention
* Inability to understand French
* Patient refusal to participate in the study and/or inability to express consent or sign the informed consent form
* Patient subject to legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-02 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the predictive value of atrial heart disease characterized by multiparametric MRI (late enhancement fibrosis, atrial strain, and exploratory 4D flow parameters) for the recurrence of atrial fibrillation documented by Implantable Loop Recorder. | through study completion, an average of 12 months
  Recurrence of atrial fibrillation, defined as an episode lasting ≥ 30 seconds documented by the Implantable Loop Recorder (ILR) implanted preoperatively and recorded during the 12-month follow-up period.

SECONDARY OUTCOMES:
Evaluate the link between atrial heart disease characterized by MRI (fibrosis, strain, 4D flow) and the occurrence of postoperative atrial fibrillation (POAF) during the first week following coronary artery bypass grafting. | through the first postoperative week
  POAF will be defined as an episode of AF ≥ 30 seconds, detected by the preoperatively implanted ILR and recorded during the first postoperative week.
Correlate MRI parameters of atrial remodeling with histological assessment of fibrosis on intraoperative atrial biopsy | through the first postoperative week
  Percentage of histological fibrosis. Analysis of atrial fibrosis using Masson's trichrome staining on intraoperative atrial biopsy (normal threshold ≤ 10%). The objective is to establish a correlation between histological data and MRI parameters.
Exploring the value of atrial hemodynamic parameters obtained by 4D flow MRI (vorticity, intra-atrial velocities) as predictive markers of atrial fibrillation | Before the surgery
  measurement of intra-auricular blood flow using 4D-flow MRI, including velocities (cm/s), flow volumes (mL/s or mL), and vorticity indices (s-¹)
To study the association between serum inflammatory biomarkers (CRP, IL-1, TNF-α) and Atrial Fibrillation recurrence. | before the surgery
  Preoperative measurement of pro-inflammatory cytokines (IL-1, TNF-α, CRP).
Determine the impact of atrial fibrillation recurrence documented by ILR on the occurrence of major cardiovascular events | through study completion, an average of 12 months
  Number of ischemic strokes, hospitalizations for heart failure, cardiovascular deaths occurring within one year of surgery, and all-cause deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste GUICHARD, MD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No